CLINICAL TRIAL: NCT05022108
Title: Alpha-Bisabolol Gel With Antihistamine Action
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Adriana Rodrigues dos Anjos Mendonça, Principal Investigator, Universidade do Vale do Sapucai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Antihistamine
Record Dates: First submitted 2021-06-12; First posted 2021-08-26 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Wounds and Injuries
Keywords: Histamine Antagonists; Phytotherapy; Wounds and injuries; Bites and Stings; Plant Oils
MeSH Terms: conditions — Wounds and Injuries; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Antihistamine test (Experimental): The forearm was sensitized at four points (A, B, C and D). Point A: positive control sensitized with a drop of histamine at a concentration of 10 mg / Ml. Point B: histamine was applied and immediately after, the alpha bisabolol gel with a concentration of 0.5%. Point C: histamine and gel with 2.5% alpha-bisabolol were applied. Point D was sensitized with a drop of histamine and 5.0% alpha-bisabolol gel. The test reading at each point occurred 15 minutes after the procedure.
  Interventions: Biological: Alpha bisabolol gel

INTERVENTIONS:
Biological: Alpha bisabolol gel — Using alpha bisabolol gel with a concentration of 0.5%, 2,5% or 5% to treat sensitized area with histamine.

SUMMARY:
It will be developed and evaluated the antihistamine potential of a gel containing alpha-bisabolol. Method: Interventional and cross-sectional study, with convenience sampling, conducted with 20 volunteers. The forearm will be sensitized at four points (A, B, C and D). Point A: positive control will be sensitized with a drop of histamine at a concentration of 10 mg / Ml. Point B: histamine will apply and immediately after, the alpha bisabolol gel with a concentration of 0.5%. Point C: histamine and gel with 2.5% alpha-bisabolol will apply. Point D will be sensitized with a drop of histamine and 5.0% alpha-bisabolol gel. The test reading at each point will occur 15 minutes after the procedure. For the analysis of the results, the T Test will be applied.

DETAILED DESCRIPTION:
Context:. Phytotherapy has been widely used to treat health with a prophylactic, curative and palliative purpose due to its easy access and low cost when compared to other available drug forms. Some plant species have antiallergic and anti-inflammatory properties that can be used to help contain signs and damage in allergic reactions, triggered mainly by histamine such as: pain, redness, heat and edema. Alpha-bisabolol, extracted from Candeia, has several applications in the treatment of illnesses, however, there are no studies on the therapeutic potential for antihistamine. Objective: To develop and evaluate the antihistamine potential of a gel containing alpha-bisabolol. Method: Pilot study, interventional, cross-sectional study, with convenience sampling, conducted with 20 volunteers. The forearm will be sensitized at four points (A, B, C and D). Point A: positive control sensitized with a drop of histamine at a concentration of 10 mg / Ml. Point B: histamine will be applied and immediately after, the alpha bisabolol gel with a concentration of 0.5%. Point C: histamine and gel with 2.5% alpha-bisabolol will be applied. Point D will be sensitized with a drop of histamine and 5.0% alpha-bisabolol gel. The test reading at each point will occur 15 minutes after the procedure. For the analysis of the results, the T Test will be applied.

ELIGIBILITY:
Inclusion Criteria:

* participants without allergy-related diseases, non-pregnant women and who agreed to cooperate in carrying out the research by signing the consent form aged between 18 and 60 years of both sexes.

Exclusion Criteria:

* participants who had a history of previous anaphylaxis, extensive dermatitis, use of antihistamines, colds or steroids.
* participants who had a negative reaction to histamine and/or withdrew their consent at any stage of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Measure of the area (cm2) sensitized with histamine only | 15 minutes
  Positive control sensitized with a drop of histamine at a concentration of 10 mg / Ml, and after 15 minutes the area sensitized will be measure
Measure of the area (cm2) sensitized by histamine treated with 0,5% Alpha bisabolol | 15 minutes
  Histamine will be applied and immediately after, the alpha bisabolol gel with a concentration of 0.5%, and after 15 minutes the area sensitized will be measure
Measure of the area sensitized by histamine treated with 2,5% Alpha bisabolol | 15 minutes
  Histamine will be applied and immediately after, the alpha bisabolol gel with a concentration of 2,5% will applied, and after 15 minutes the area sensitized will be measure
Measure of the area (cm2) sensitized by histamine treated with 5% Alpha bisabolol | 15 minutes
  It will be sensitized with a drop of histamine and immediately with 5.0% alpha-bisabolol gel, and after 15 minutes the area sensitized will be measure

CONTACTS AND LOCATIONS:
Overall Officials: Adriana R dos Anjos Mendonça, PhD, Principal Investigator — Vale do Sapucaí University
Locations (1):
- Vale do Sapucaí University, Pouso Alegre, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No